CLINICAL TRIAL: NCT06181253
Title: The Impact of Prehabilitation Measures on Postoperative Outcomes
Brief Title: The Impact of Prehabilitation
Acronym: Prehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-42768
Record Dates: First submitted 2023-12-05; First posted 2023-12-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Post Operative Complications
Keywords: Prehabilitation; Patient video education; Instructional walking video; 6 minute Walking test; Patient texting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): Watch a video created by the investigators, discussing exercise prior to surgery, receive text message reminders to begin exercise before surgery, and take walking tests before and after surgery.
  Interventions: Other: Preoperative education; Behavioral: Moderate aerobic exercise; Other: Text messages; Behavioral: Pedometer
- Control group (No Intervention): Receive the usual preoperative and post operative care and they will be provided a pedometer.

INTERVENTIONS:
Other: Preoperative education — The intervention will be an instructional video describing proper walking technique particularly up flights of stairs for patients to do at home. This will be shown at preoperative surgical clinic and will be available for access at home from patient's cell phones. The video is currently in production at BMC. Additionally, text reminders will be sent daily to remind patients to walk at home.
  Arms: Prehabilitation group
Behavioral: Moderate aerobic exercise — Participants will be encouraged to compete 140-150 minutes of moderate aerobic exercise per week- achieved by two walking sessions per day 10-11 minutes in length (realistic/achievable goal)
  Arms: Prehabilitation group
Other: Text messages — Text reminders will be sent daily to remind patients to walk at home.
  Arms: Prehabilitation group
Behavioral: Pedometer — Participants will be encouraged to walk 10,000 steps daily which will be tracked with a pedometer
  Arms: Prehabilitation group

SUMMARY:
While numerous studies have assessed the promising impacts of prehabilitation, there is a lack of prehabilitation research within lower socioeconomic patient populations. Often for prehabilitation studies, patients are heavily involved in full scale exercise and nutrition programs weeks before the scheduled procedure. In underserved populations, programs such as these are often not feasible due to lack of transport, resources, and other barriers to healthcare. The investigators seek to evaluate the effectiveness of inexpensive interventions in lower socioeconomic populations.

The investigators hypothesize that barriers to prehabilitation are environmental and that prehabilitation interventions tailored for lower socioeconomic (SES) populations will improve time to discharge, mobility, and in turn, readmission rates.

The participants for this clinical trial will be seen four times: initially at the preoperative surgical clinic (6-8 weeks prior to surgery), 1-2 days preop at a pre-procedure clinic, postoperative in the inpatient setting (as soon as the participant is able to ambulate during their hospital stay), and in the postoperative surgical clinic at the postoperative visit. Patients will be within the general surgery, colorectal, and surgical oncology departments at Boston Medical Center (BMC).

The anticipated sample size is 60 participants (30 in the intervention/prehabilitation arm and 30 in the control/usual care arm). Participants in the intervention arm will participate in a mobility and step tracking intervention aimed at improving postoperative outcomes. The control group will follow routine standard of care at BMC for preoperative and postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients within general surgery, colorectal, and surgical oncology departments at Boston Medical Center.
* English or Spanish speaking
* Able to ambulate without cane, walker, wheelchair
* Surgery scheduled within 4-8 weeks
* Must have cell phone with internet access and text message capabilities
* JH-HLM score of 6

Exclusion Criteria:

* Limited/non readers (less than 5th grade reading level), assessed via comprehension of consent materials

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Baseline 6 minute walking test (6MWT) | Baseline (preoperatively)
  The 6MWT is an exercise test that measure patient endurance and aerobic capacity. Participants will walk while attached to pulse oximetry for 6 minutes and total distance walked will be recorded. The higher a person's score, the better their exercise tolerance.
Postoperative 6 minute walking test (6MWT) | Postoperative, 24-48 hours after surgery
  The 6MWT is an exercise test that measure patient endurance and aerobic capacity. Participants will walk while attached to pulse oximetry for 6 minutes and total distance walked will be recorded. The higher a person's score, the better their exercise tolerance.
Baseline Activity Measure for Post Acute Care (AMPAC) | Baseline (preoperatively)
  This tool aims to assess a patient's physical function status as it relates to activities of daily living as a brief questionnaire. Questions assess ability to perform activities such as dressing and ambulating.Known as "6-Clicks" due to being composed of six scored patient activity questions, a patient's "6-Clicks" score falls on a 6- to 24-point scale where a score of 6 represents total functional impairment and a score of 24 represents total absence of impairment.
Postoperative Activity Measure for Post Acute Care (AMPAC) | Postoperative, 24-48 hours after surgery
  This tool aims to assess a patient's physical function status as it relates to activities of daily living as a brief questionnaire. Questions assess ability to perform activities such as dressing and ambulating.Known as "6-Clicks" due to being composed of six scored patient activity questions, a patient's "6-Clicks" score falls on a 6- to 24-point scale where a score of 6 represents total functional impairment and a score of 24 represents total absence of impairment.
Baseline Frailty Scoring | Baseline (preoperatively)
  Clinical frailty score is a 9 point scale used to assess frailty in patients. A score of 1 indicates "Very Fit", 2 indicates "Fit", and so on. A frailty score of 9 indicates terminally ill. The higher the frailty score, the more frail a patient is considered. Clinicians use their best judgement given a variety of patient factors including physical fitness, motivation, and medical comorbidities
Postoperative Frailty Scoring | Postoperative, 24-48 hours after surgery
  Clinical frailty score is a 9 point scale used to assess frailty in patients. A score of 1 indicates "Very Fit", 2 indicates "Fit", and so on. A frailty score of 9 indicates terminally ill. The higher the frailty score, the more frail a patient is considered. Clinicians use their best judgement given a variety of patient factors including physical fitness, motivation, and medical comorbidities.
Baseline John's Hopkins Highest Level of Mobility (JH-HLM) Scale | Baseline (preoperatively)
  The JH-HLM is an ordinal scale for documenting a patient's highest observed level of activity in the bed, chair, standing, and walking. It has a range from 1 to 8 where lying in bed (score = 1) to ambulating >250 feet (score = 8). HIgher scores indicate greater mobility.
Postoperative John's Hopkins Highest Level of Mobility (JH-HLM) Scale | Postoperative, 24-48 hours after surgery
  The JH-HLM is an ordinal scale for documenting a patient's highest observed level of activity in the bed, chair, standing, and walking. It has a range from 1 to 8 where lying in bed (score = 1) to ambulating >250 feet (score = 8). HIgher scores indicate greater mobility.
Baseline Veterans Rand 12 (VR-12) Item Health Survey | Baseline (preoperatively)
  The VR-12 is a patient reported outcome measure that aims to assess patients health related qualify of life as it relates to their physical and mental health.The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS and MCS are both 50 points.
Postoperative Veterans Rand 12 (VR-12) Item Health Survey | Postoperative, 24-48 hours after surgery
  The VR-12 is a patient reported outcome measure that aims to assess patients health related qualify of life as it relates to their physical and mental health.The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS and MCS are both 50 points.
Adherence to mobility intervention assessed by text survey data | 8 weeks
  Participants will be asked daily regarding home activity level (minutes of walking per day) as a measure of adherence to prehabilitation walking program.
Adherence to mobility intervention assessed by pedometer step count | 8 weeks
  Participants will be asked daily about their pedometer step count as a measure of adherence to prehabilitation walking program.

SECONDARY OUTCOMES:
Readmission rate | 8 weeks
  Through chart review, the participants readmission rate back into the hospital (postoperatively) will be compared between the intervention and control group.
Length of hospital stay | 6-8 weeks
  The number of days participants are hospitalized will be abstracted from the participants medical records.
Complications from surgery | 2 months post surgery
  Through chart review, the rate of complications will be compared intervention and control group. Complications comprise of: infection of surgical site, hemorrhage, deep vein thrombosis and pulmonary embolism, pulmonary complications (ie. atelectasis, pneumonia), and death.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Spence, MD, Principal Investigator — Boston Medical Center, Anesthesiology Department
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No